CLINICAL TRIAL: NCT06923111
Title: A Comparative Observational Study to Evaluate the Safety and Effectiveness of Xromi (Hydroxycarbamide Oral Solution 100mg/ml) for the Prevention of Vaso-occlusive Complications of Sickle Cell Disease in Children Under 2 Years of Age.
Brief Title: PASS of Xromi Comparing Safety and Effectiveness in Children Under 2 Years With Sickle Cell Disease [PRECISE PASS]
Acronym: PRECISE
Status: Recruiting | Type: Observational
Sponsor: Nova Laboratories Limited (Industry)
Collaborators: OXON Epidemiology (Industry)
Responsible Party: Sponsor
Other Study IDs: NOVDD-001; EUPAS1000000076 (Other: HMA-EMA RWD Catalogues); CHIL 62837 (Other: NIHR CPMS); 334976 (Other: HRA IRAS)
Record Dates: First submitted 2025-04-03; First posted 2025-04-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxyurea; liquid formulation; HbS Disease; Hemoglobin S Disease; Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Disorders; Sickling Disorder Due to Hemoglobin S; Xromi; Hydroxycarbamide; paediatric; children; hemaglobinopathy in children; hemoglobinopathy; paediatric formuation
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies | interventions — Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Exposure Cohort: Children with SCD aged 9 months to under 2 years of age who are newly prescribed Xromi®, will be identified prospectively. These participants will be followed up for 24 months from their index date, regardless of whether they continue treatment with Xromi®, discontinue all hydroxycarbamide treatment, or switch to another formulation of hydroxycarbamide. The decision to prescribe Xromi® will be made solely by the physician independently of the study, as part of standard care.
  -
  Interventions: Drug: Xromi
- Retrospective Comparator Cohort: Children with SCD and naïve to any hydroxycarbamide formulation at the index date. These participants will be identified retrospectively using the data from the last 10 years up to the date Xromi® was first used in children from 9 months to under 2 years of age at each individual site. The 24-month follow-up will be retrospective from the date they are matched to the exposed participant, irrespective of whether they start on any formulation of hydroxycarbamide during the follow-up.

INTERVENTIONS:
Drug: Xromi — Xromi is indicated for the prevention of vaso-occlusive complications of Sickle Cell Disease in patients over 9 months of age as part of standard clinical practice
  Other Names: hydroxycarbamide oral solution 100mg/ml; liquid hydroxyurea; LO1XX05
  Groups: Prospective Exposure Cohort

SUMMARY:
This post-authorisation safety and efficacy study (PRECISE PASS) evaluates the use of Xromi® (hydroxycarbamide 100 mg/mL oral solution) in children aged 9 months to under 2 years with sickle cell disease (SCD).

The objective is to assess the safety profile and clinical effectiveness of Xromi® under routine clinical conditions. The study includes a prospective cohort of Xromi®-treated patients and a matched retrospective comparator cohort of untreated patients. Participants will be followed for 24 months from treatment initiation or matched index date.

DETAILED DESCRIPTION:
The PRECISE study is a combined Post-Authorisation Safety Study (PASS) (Category 3) and a Post-Authorisation Efficacy Study that aims to provide data on the safety and effectiveness of hydroxycarbamide 100mg/ml oral solution (Xromi ®) administered prospectively to children under 2 years of age, over a follow-up period of 24 months compared to matched retrospective comparators who were treatment naïve.

This is a non-interventional, matched cohort study involving children with SCD aged 9 to under 24 months. The study comprises two groups:

* A prospective Xromi®-exposed cohort, enrolled at the time of treatment initiation and followed for 24 months.
* A retrospective comparator cohort, matched 2:1 by site, age, and β-globin genotype, identified from clinical records of children not treated with hydroxycarbamide at the index date.

The primary objective is to compare the incidence of adverse events of special interest (AESIs) between the two cohorts. Secondary analyses will assess the comparative effectiveness of Xromi® on clinical events, laboratory parameters, and physiological assessments. Exploratory analyses will examine treatment-related safety and effectiveness by dose, subgroups, and exposure to hydroxycarbamide during follow-up.

Data will be sourced from routine clinical practice through chart reviews and follow-up visits. No study-specific interventions will be introduced. The study is planned across specialist sites in the UK and Germany, with potential expansion to other European countries if recruitment targets require.

ELIGIBILITY:
Prospective Exposure Cohort

* Inclusion criteria:

  * Aged from 9 months to under 2 years at the index date.
  * Diagnosis of SCD.
  * Known β-globin genotype at the index date.
  * Prescribed Xromi® for the prevention of complications of SCD.
  * Parent(s) (or a legal representative(s)) provides written informed consent to participate in the study, unless there is a waiver, non-opposition, or blanket written informed consent by the parent for research studies.
* Exclusion criteria:

  * Previous use of hydroxycarbamide of any formulation before the index date.
  * Receiving regular blood transfusions (occurring every 8 weeks or more frequently) at the index date.
  * Known hypersensitivity to any of the excipients of Xromi® at the index date.
  * Contraindications to the drug at the index date: severe hepatic impairment (Child-Pugh classification C); severe renal impairment (creatinine clearance: CrCl <30 ml/min); presence of at least one of the following: Absolute neutrophil count (ANC) < 1.0 x 10^9/L, absolute reticulocyte count (ARC) <80 x 10^9/L, platelets <80 x 10^9/L.
  * Participating in another clinical study of an investigational medicinal product (IMP) at the index date.
  * Anti-retroviral medicinal products for human immunodeficiency virus (HIV) at the index date.
  * Active malignancy at the index date.

Participants in the prospective exposure cohort who are prescribed Xromi® but do not initiate treatment will be excluded from the dataset.

Retrospective Comparator cohort

* Inclusion criteria:

  * Aged from 9 months to under 2 years at the index date.
  * Diagnosis of SCD.
  * Known β-globin genotype.
  * Matched to an exposed participant.
  * Parent(s) (or a legal representative(s)) provides written informed consent to participate in the study, unless there is a waiver, non-opposition, or blanket written informed consent by the parent for research studies.
* Exclusion criteria:

  * Use of hydroxycarbamide of any formulation before or at the index date.
  * Receiving regular blood transfusions (occurring every 8 weeks or more frequently) at the index date.
  * Presence at the index date of any of the following: severe hepatic impairment (Child-Pugh classification C); severe renal impairment (CrCl <30 ml/min); presence of at least one of the following: ANC < 1.0 x 10^9/L, ARC < 80 x 10^9/L, platelets < 80 x 10^9/L).
  * Participating in another clinical study of an IMP at the index date.
  * Anti-retroviral medicinal products for HIV at the index date.
  * Active malignancy at the index date.

Ages: 9 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will consist of children with SCD who meet all the inclusion criteria and none of the exclusion criteria.
  Identification of participants will be conducted as follows:
  * Prospective exposure cohort: Potential participants will be identified as they attend the participating sites where eligibility criteria will be assessed prior to initiation with Xromi.
  * Retrospective comparator cohort: Potential participants will be selected from clinical chart review for hydroxycarbamide naive children that could be matched to prospective participants.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
AESI - Myelosuppression (Neutropenia) | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Myelosuppression protocol definition of neutropenia is ANC <1.0 x 10^9/L
AESI - Myelosuppression (Reticulocytopenia) | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Myelosuppression protocol definition of reticulocytopenia is ARC <80 x 10^9/L, unless Hb >90 g/L,
AESI - Myelosuppression (Thrombocytopenia) | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Myelosuppression protocol definition of thrombocytopenia defined as platelets <80 x 10^9/L.
AESI - Myelosuppression (Anaemia) | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Myelosuppression protocol definition of anaemia defined as Hb <45 g/L.
AESI - Abnormal Weight Gain | Baseline to 24 months
  Weight (kg) Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort and standard care guidelines
AESI - Abnormal Weight Loss | Baseline to 24 months
  Weight (kg) Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort and standard care guidelines
AESI - Increase in Hepatic Enzyme (ALT) | Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort and normal laboratory ranges. Defined as an increase in hepatic enzyme Alanine transaminase (ALT) increased (U/L)
AESI - Increase in Hepatic Enzyme (AST) | Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort and normal laboratory ranges. Defined as an increase in hepatic enzyme Aspartate transaminase (AST) increased (U/L)
AESI - Alopecia | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in study protocol as presence of alopecia (a skin and subcutaneous tissue disorder).
AESI - Other Hair Loss | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in study protocol as presence of other hair loss (a skin and subcutaneous tissue disorder).
AESI - Skin Hyperpigmentation | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in study protocol as presence of skin hyperpigmentation, including oral and nail hyperpigmentation.(a skin and subcutaneous tissue disorder).
AESI - Rash | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in study protocol as presence of a rash (a skin and subcutaneous tissue disorder).
AESI - Skin Ulcers | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in study protocol as presence of skin ulcer, including leg ulcer (a skin and subcutaneous tissue disorder).
AESI - Growth Retardation | Pre-baseline, Baseline to 24 months
  height/length (cm) Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort and standard care guidelines (as a drop of 2 or more centiles on growth charts over time).
AESI - Bacterial Infection | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in the protocol as a proven or treated bacterial infection.
AESI - Viral Infection | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in the protocol as a proven or treated viral infection.
AESI - Fungal Infection | Pre-baseline, Baseline to 24 months
  Incidence of adverse events of special interest (AESIs) in children who have SCD and are treated with Xromi®, in comparison to a retrospective comparator cohort. Defined in the protocol as a proven or treated fungal infection.

SECONDARY OUTCOMES:
Other Adverse Events | Baseline to 24 months
  Occurrence of other adverse events (AE), adverse reactions (AR) and serious adverse events (SAE) or serious adverse reactions (SAR) will be collected during follow-up.
Painful Vaso-occlusive Crisis (VOC) | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  - VOC events will include dactylitis.
Acute Chest Syndrome (ACS) | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Splenomegaly | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event Splenomegaly will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Priapism | Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Hepatobiliary disorder | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Splenic Sequestration Crisis | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Surgery | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  Defined in the protocol as any surgery that is planned, emergency, or due to pre-existing conditions e.g. SCD.
Blood Transfusion | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Cerebrovascular accident | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  The protocol definition includes silent stroke
Abnormal or Conditional TCD | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  - Transcranial Doppler Scan (TCD)
Hospitalisations for SCD | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  The reason for hospitalisation and duration will be collected.
Non-hospitalised Visit for SCD | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
  Protocol definition includes Emergency department (ED) visits/treatment centres/paediatric ward/day unit attendances for SCD
Other Clinical Events | Pre-baseline, Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator to compare the Effectiveness of Xromi®.
Other Event - Death | Baseline to 24 months
  Occurrence of the clinical event will be collected during follow-up in both cohorts by the investigator. Protocol definition includes any death occurring in the study both related and un-related to Xromi treatment
Haemoglobin (Hb) | Pre-baseline, Baseline to 24 months
  (g/L) or (g/dl) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Foetal Haemoglobin (HbF) | Pre-baseline, Baseline to 24 months
  (%) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Haemoglobin Fractions | Pre-baseline, Baseline to 24 months
  (%) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
  - Haemoglobinopathy screen results including: HbS, HbA, HbA2, HbC
Absolute Neutrophil Count (ANC) | Pre-baseline, Baseline to 24 months
  (10^9/L or /nL) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Absolute Reticulocyte Count (ARC) | Pre-baseline, Baseline to 24 months
  (10^9/L or /nL) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Platelet Count | Pre-baseline, Baseline to 24 months
  (10^9/L or /nL) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
White Blood Cell Count (WBC) | Pre-baseline, Baseline to 24 months
  (10^9/L or /nL) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Mean Corpuscular Volume (MCV) | Pre-baseline, Baseline to 24 months
  (fl) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Mean Corpuscular Haemoglobin (MCH) | Pre-baseline, Baseline to 24 months
  (pg) Haematological Parameter. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Ferritin | Pre-baseline, Baseline to 24 months
  (µg/L) Iron Profile. Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Transferrin Saturation | Pre-baseline, Baseline to 24 months
  (%) Iron Profile. Iron binding saturation or transferrin saturation.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Alanine Transaminase (ALT) | Pre-baseline, Baseline to 24 months
  (U/L) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Alkaline Phosphatase (ALP) | Pre-baseline, Baseline to 24 months
  (U/L) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Aspartate Transaminase (AST) | Pre-baseline, Baseline to 24 months
  (U/L) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Total Bilirubin | Pre-baseline, Baseline to 24 months
  (µmol/L or mg/dl) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Lactate Dehydrogenase | Pre-baseline, Baseline to 24 months
  (U/L) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Gamma-Glutamyl Transferase (GGT) | Pre-baseline, Baseline to 24 months
  (U/L) Liver Function tests.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Serum Creatinine | Pre-baseline, Baseline to 24 months
  (µmol/L or mg/dl) Renal function test.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Estimated Glomular Filtration Rate (eGFR) | Pre-baseline, Baseline to 24 months
  (ml/min/1.73m^2) Renal function test. Calculated value, Interpreted in line with UK CKD guidelines from creatinine values.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Albumin-Creatinine Ratio (ACR) | Pre-baseline, Baseline to 24 months
  (Calculated value). Renal function test.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Liver Size | Pre-baseline, Baseline to 24 months
  (cm) from costal margin. Physiological Assessment.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Spleen Size | Pre-baseline, Baseline to 24 months
  (cm) from costal margin. Physiological Assessment.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.
Maximum Time Averaged Mean Velocity (TAMV) | Pre-baseline, Baseline to 24 months
  (cm/s) Cardiovascular function, assessed using transcranial doppler scan velocities.
  Results and dates of laboratory tests and physiological assessments will be collected, whenever available. At baseline, the most recent results, prior to Xromi® initiation in the prospective exposure cohort, will be collected. Results from laboratory tests and physiological assessments conducted during follow-up will also be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Hussain Dr Mulla, PhD, Study Director — Nova Laboratories Ltd.; Sara Dr Trompeter, MD, Principal Investigator — University College London Hospitals
Locations (5):
- United Kingdom (5):
  - Basildon University Hospital, Basildon, Essex
  - Noah's Ark Children's Hospital for Wales, Cardiff, Leicestershire
  - University College London Hospital, London, North London
  - The Royal London Hospital, London, Whitechapel
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The study has been registered on a public database HMA-EMA RWD Catalogues and the study protocol has been shared publicly (EUPAS1000000076).
  Study publication of aggregated outcome results on Clinical trials.gov and in Multi-centre study publication in relevant medical journal.
  Investigators:
  All Investigators will be provided with their individual participant data at the end of the study as eCRFs.
  Regulatory Authorities:
  The study protocol was shared with the EMA and MHRA. The draft SAP was shared with the EMA during initial review of the study protocol prior to study initiation.
  CSR will be made available to the EMA and MHRA at the end of the study.
Supporting Information: Study Protocol
Time Frame: March 2025 - upto 25 years from end of study.
Access Criteria: Publicly accessible study protocol via the HMA-EMA RWD Catalogues and the study protocol has been shared publicly (EUPAS1000000076) Publicly accessible aggregated study results via ClinicalTrials.Gov.

REFERENCES:
- [Background] Rankine-Mullings A, Keenan R, Chakravorty S, Inusa B, Telfer P, Velangi M, Ware RE, Moss JJ, Lloyd AL, Edwards S, Mulla H. Efficacy, safety, and pharmacokinetics of a new, ready-to-use, liquid hydroxyurea in children with sickle cell anemia. Blood Adv. 2023 Aug 22;7(16):4319-4322. doi: 10.1182/bloodadvances.2023010099. No abstract available. PMID 37171600
- [Background] Thompson BW, Miller ST, Rogers ZR, Rees RC, Ware RE, Waclawiw MA, Iyer RV, Casella JF, Luchtman-Jones L, Rana S, Thornburg CD, Kalpatthi RV, Barredo JC, Brown RC, Sarnaik S, Howard TH, Luck L, Wang WC. The pediatric hydroxyurea phase III clinical trial (BABY HUG): challenges of study design. Pediatr Blood Cancer. 2010 Feb;54(2):250-5. doi: 10.1002/pbc.22269. PMID 19731330